CLINICAL TRIAL: NCT07267169
Title: Lipopolysaccharide Adsorption (Efferon LPS) in Patients With Acute Pancreatitis
Brief Title: Efferon LPS Hemoadsorption in Patients With Acute Pancreatitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efferon JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: efferon-lps-2025-02
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Pancreatitis, Acute
Keywords: acute pancreatitis; hemoperfusion
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Intervention Model Description: Allocation of patients into groups will be done by stratified 1:1 randomisation.
  Stratification factors will include the Sequential Organ Failure Assessment (SOFA) score, Computed Tomography Severity Index (CTSI), and blood lactate levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline therapy+ HF/HDF (No Intervention): Basic therapy - which is the routine practice of an institution for the treatment of patients with uninfected acute pancreatitis in combination with hemofiltration (HF) or hemodiafiltration (HDF) procedures.
- Baseline therapy + HF/HDF + Efferon LPS (Experimental): Patients will receive basic therapy (routine practice of an institution for the treatment of patients with uninfected acute pancreatitis), hemofiltration or hemodiafiltration procedures in combination with hemoadsorption therapy (Efferon LPS).
  Interventions: Device: Efferon LPS

INTERVENTIONS:
Device: Efferon LPS — Efferon LPS, a medical device, which is a single-use cartridge filled with a polymeric adsorbent that selectively adsorbs endotoxin via surface-immobilized ligand and excessive cytokines via its intrinsic porosity.
  Efferon LPS will be administered in combination with either hemofiltration (HF) or hemodiafiltration (HDF). The choice between HF and HDF will be made by the investigator, based on the individual clinical situation.The therapy will be initiated within the first 24 hours after ICU admission and within 8 hours after patient enrollment.
  Arms: Baseline therapy + HF/HDF + Efferon LPS

SUMMARY:
The goal of the study is to evaluate the safety and efficacy of multimodal (cytokine and lipopolysaccharide) hemoperfusion using the Efferon® LPS device in combination with hemofiltration (HF) / hemodiafiltration (HDF), with the goal of reducing the severity of organ dysfunction (measured by SOFA score) in patients with acute pancreatitis.

Participants will be assigned to two groups for comparison: a control group receiving baseline therapy with HF/HDF, and a treatment group receiving baseline therapy in combination with HF/HDF and Efferon® LPS hemoadsorption.The therapy will be initiated within the first 24 hours after ICU admission and within 8 hours after patient enrollment.

DETAILED DESCRIPTION:
Acute pancreatitis remains a life-threatening disorder with a considerable risk of unfavorable outcomes. In patients with severe acute pancreatitis (SAP), hospital mortality ranges from 16% to 20% and may rise to 60% in cases complicated by multiple organ dysfunction (MOD). Progressive MOD, arising from systemic inflammatory response syndrome (SIRS), represents the principal cause of early death. Recently, extracorporeal blood purification techniques, including hemoperfusion, have emerged as valuable adjuncts to intensive care, providing opportunities to correct derangements in homeostasis.

In recent years, extracorporeal blood purification methods, including hemoperfusion, have become one of the components of intensive care, allowing for correction of homeostatic parameters.

The Efferon® LPS device was originally developed for use in sepsis, utilizing its ability to effectively target both primary and secondary inflammatory mediators. However, this approach also has significant potential for the treatment of acute pancreatitis, a condition characterized by a similarly complex inflammatory response.

The goal of the study is to evaluate the safety and efficacy of multimodal (cytokine and lipopolysaccharide) hemoperfusion using the Efferon® LPS device in combination with hemofiltration/hemodiafiltration, with the goal of reducing the severity of organ dysfunction in patients with acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* ≤ 5 days from the onset of acute pancreatitis
* Acute pancreatitis of moderate or severe according to the Atlanta classification (2012)
* Acute pancreatitis confirmed by tomography. Modified CTSI Pancreatitis Severity Index Score ≥ 4 points
* APACHE II > 8
* ≥ 2 points on the Sequential Organ Failure Assessment (SOFA) scale and/or ≥ 2 criteria of Systemic Inflammatory Response Syndrome (SIRS):
* Body temperature ≥ 38 °C or ≤ 36 °C
* Heart rate ≥ 90/min
* Respiratory rate ≥ 20/min or hyperventilation with PaCO₂ ≤ 32 mmHg
* Leukocytosis (≥ 12,000/μl) or leukopenia (≤ 4,000/μl) or left shift of leukocyte formula

Exclusion Criteria:

* SOFA score > 12 points
* Presence of an uncontrolled surgical infection focus
* Development of septic complications - signs of infection
* Acute pancreatitis as an exacerbation of chronic pancreatitis
* Blood triglyceride level > 1000 mg/dL (11.2 mmol/L)
* Liver cirrhosis (> 6 points by Child-Pugh classification)
* Unresolved biliary hypertension syndrome
* BMI ≥ 40
* Dementia
* Chronic kidney disease stage 4-5
* Acute pulmonary embolism confirmed by CT
* Acute myocardial infarction within the last 4 weeks
* Acute cerebrovascular accident
* Severe congestive heart failure
* Uncontrolled bleeding (acute blood loss within the last 24 hours)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
SOFA score | 1-7 days
  The Sequential Organ Failure Assessment (SOFA) score is equal to the sum of six indicators. The higher the score, the greater the insufficiency of the system being assessed. The higher the overall score, the greater the degree of multiorgan dysfunction. Violation of the function of each organ (system) is assessed separately in dynamics against the background of intensive therapy. With a score of no more than 12, multiple organ dysfunctions are assumed, 13-17 points indicate the transition of dysfunction to insufficiency, a score of about 24 indicates a high probability of death. The lower the SOFA score, the less pronounced organ failure and the better the patient's survival prognosis.

SECONDARY OUTCOMES:
Vasopressor free days | 1-14 days
  * Vasopressor free days = 0 if subject dies within 14 days of starting vasopressor support.
  * Vasopressor free days = 14 - x if vasopressor support is successfully discontinued x days after initiation.
  * Vasopressor free days = 0 if the subject requires vasopressor support for more than 14 days.
Horovitz oxygenation index | 1-14 days
  Value of oxygenation index (Pa02 / Fi02 (Pa).
  Oxygenation index (PaO₂/FiO₂) = arterial oxygen partial pressure (Pa02, mmHg) / the fraction of inspired oxygen (FiO2).
Cardiac index | 1-72 hours
  Cardiac index = stroke volume (mL/beat) × heart rate (beats/min) / BSA (m²)
  BSA - body surface area
Length of stay in the intensive care unit | 1-60 days
  Time (number of days) from randomization to transfer from the intensive care unit within 60 days.
Mechanical ventilation duration | 1-28 days
  * Ventilator-free days = 0 if subject dies within 28 days of mechanical ventilation.
  * Ventilator-free days = 28 - x if successfully liberated from ventilation x days after initiation.
  * Ventilator-free days = 0 if the subject is mechanically ventilated for >28 days.
Renal replacement therapy (RRT) duration | 1-28 days
  * RRT-free days = 0 if the subject dies within 28 days of starting renal replacement therapy.
  * RRT-free days = 28 - x if RRT is successfully discontinued x days after initiation.
  * RRT-free days = 0 if the subject requires RRT for more than 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Kiselev, PhD, MD, Principal Investigator — N. V. Sklifosovsky Moscow Research Institute of Emergency
Locations (8):
- Russia (8):
  - Republican Clinical Hospital of the Ministry of Health of the Republic of Tatarstan, Kazan'
  - State Clinical Hospital "Regional Clinical Hospital No 2" of the Ministry of Healthcare of Krasnodar Territory, Krasnodar
  - V.P. Demikhov City Clinical Hospital No. 68, Moscow
  - S.S. Yudin City Clinical Hospital, Moscow
  - N.I. Pirogov City Clinical Hospital No. 1, Moscow
  - N.V. Sklifosovsky Research Institute for Emergency Medicine, Moscow
  - Perm regional clinical hospital, Perm
  - North-Western district scientific and clinical center named after L. G. Sokolov Federal Medical and Biological Agency, Saint Petersburg